CLINICAL TRIAL: NCT05306587
Title: Daratumumab Provided at Home Experience: An Open, Single-center, Mixed-method Project Initiated on Behalf of Odense University Hospital
Brief Title: Daratumumab Provided at Home Experience An Open, Single-center, Mixed-method Project.
Status: Completed | Type: Observational
Sponsor: Thomas Lund (Other)
Responsible Party: Sponsor-Investigator, Thomas Lund, Principal Investigator, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: DAPHNE
Record Dates: First submitted 2021-12-06; First posted 2022-04-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Multiple Myeloma: 40 patients with Multiple Myeloma in Department of Hematology at Odense University Hospital, Denmark
  Interventions: Drug: Darzalex

INTERVENTIONS:
Drug: Darzalex — Investigate the home administration of Darzalex SC reported by both patients and healthcare professionals compared to the hospital administration setting.
  Other Names: Daratumumab

SUMMARY:
Multiple myeloma (MM) is the second most common hematological disease in Denmark with an incidence of approximately 350 diagnosed cases per year. There is no curative treatment yet, but usually the disease is very sensitive to treatment, and patients have periods of varying length, where they do not require treatment. Thus the prognosis for MM has improved over recent years, and the rate of survival has been extended for both younger and elderly patients. With the increasing specialization and centralization that will occur in the coming years, some patients will have very long transport times to the hospital. When patients go to the hospital only to receive their anticancer therapy, their visits are relatively short and the amount of time spend on transportation might appear disproportionate. The frequent hospital appointments increase the patient's exposure for bacteria and viruses which should be calculated as a potential risk. Furthermore if the patient is an active part of the labor market, it can be challenging to request freedom to hospital visits.

It is thus possible to provide the treatment at home, but it is unknown what significance it has for patients, relatives and health professionals as well as for the economy it is thus possible to provide the treatment at home, but it is unknown what significance it has for patients, relatives and health professionals as well as for the economy. The aim of this project is to investigate the home administration of Daratumumab SC reported by both patients and healthcare professionals compared to the hospital administration setting. Furthermore, this project investigates the hypothesis that the home administration of Daratumumab potentially can reduce the time associated with the administration, thereby, resulting in a socio-economic gain.

The aim for this study: We want to examine patients 'and healthcare professionals' perspectives, the organizational and the socio economic aspects of administering subcutaneous Daratumumab in their own home to patients with multiple myeloma, and to illuminate the benefits and challenges of this.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, clinical parallel mixed-methods intervention project using qualitative and quantitative data in the form of semi-structured telephone interviews, focus group interviews, time registration, registration of patients' contact with the healthcare system and PRO data. The project will both include patients already being treated with SC Daratumumab and new patients planned to start Daratumumab treatment = 40 patients in all. The patients will be included in the department of hematology Odense University Hospital as they are found eligible.

The intervention of the study is home administration of Daratumumab SC by a home nurse, thereby, changing the administration setting from a hospital setting to at home setting. The intervention with home administration will be compared to the hospital setting. The patients will function as their own controls, as treatment will be given alternately at the hospital.

Patients scheduled for Daratumumab SC at home will be phoned by a nurse from the Hematology Outpatient Clinic the day before planned administration. This procedure is chosen as that it allows the nurse to determine whether it is justifiable, for the patient to receive treatment at home. If the nurse and doctor assess that the patient is fit for home administration of Daratumumab SC, the drug will be ordered at the pharmacy to be delivered to the patient the following day. Also an electronic message will also be sent to the home nurses with an instruction to administer Daratumumab SC between 12-02 PM.

Data collection will consist of:

* Semi-structured virtual (or alternative telephone) interviews with participating patients focusing on benefits / gains versus challenges / disadvantages in regard to the actual injection, collaboration with the home nurse, delivery of medication, empowerment, and suggestions for further improvements n = 2 x 10
* Semi-structured interviews with involved home nurses n = 1 x 5.
* Focus group interview with health professionals involved at OUH at the end of the project n = 1.
* Registration of unplanned contact to the health service during the study period to account for any extra health care usage during home treatment via the app "My hospital" x 1 weekly n = 40
* Data on quality of life; EORTC custom built satisfaction questionnaire via the app "My hospital" = 5 times per patient.
* Registration of the patients evaluation of whether the use of the app "My hospital" can be useful in the future.
* Registration of patients' time used on treatment when at home or when at hospital including transport via the app "My hospital".
* Registration of the outpatient nurses' and home nurses time using the registration form via paper.
* Registration of patients general condition and possible side effects in order to clarify whether they are "fit" for treatment via the app "My hospital". This ensures that a cure that is not used is not prepared.

All Suspected Unexpected Serious Adverse Reactions (SUSARs) will be reported to the Danish National Health Authorities according national law within 7 days after awareness. Since this is not at clinical trial, but merely a collection of data during a different logistics setup, the study will be submitted to the Danish Data Protection Agency, however not to the Danish National Ethical Committee nor the Danish National Health Authorities. Due to this Adverse Reactions (AEs) will not be systematically registered or reported to the Danish national health authorities. To make sure the logistics setup is safe for all patients we will register all unplanned hospitalizations as well as all other related Serious Adverse Reactions (SAR).

Processing of personal data in the project The project is notified to the Region's Register so that it complies with the Data Protection Regulation (GDPR). All electronic data will be stored on a secure SharePoint site that can only be accessed via the project group's work computer. All physical material is stored behind double-locked doors at the project group's workplace.

ELIGIBILITY:
Inclusion Criteria:

* have relapse of MM.
* be in or have planned to start treatment with Daratumumab SC.
* be cognitively capable to assess any side effects of Daratumumab SC based on the instructions provided.
* be able and willing to register in a timetable and to participate in two semi-structured telephone interviews.
* be able to understand and speak Danish.
* be in possession of a mobile phone (for SMS tracking).

Exclusion Criteria:

- receive other anti-myeloma treatment that require hospitalization with the exception of visit 1 in all cycles with Daratumumab SC administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients planned to start treatment with SC Darzalex or patients allready in treatment with SC Darzalex.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Patients' satisfaction reported by semi-structured interviews and patient reported outcome measurements (PROM) | 01.04.2022-01.08.2024
  To analyse changes in QoL measured by EORTC IL90

SECONDARY OUTCOMES:
Examination of patients' time spend on treatment in minutes | 01.04.2022-01.08.2024
  Examination of patients' time spend on treatment in minutes through an app on a smartphone.
Examination of healthcare professionals' time spend on treatment in minutes | 01.04.2022-01.08.2024
  Examination of healthcare professionals' time spend on treatment in minutes on paper
Examination of healthcare professionals' satisfaction using focus group interview | 01.04.2022-01.08.2024
  Examination of healthcare professionals' satisfaction using focus group interview at end of study
Examination of financial perspective through calculations healthcare salaries based on time spend on treatment and transportation of medicatoin and/or patients | 01.04.2022-01.08.2024
  Examination of financial perspective through calculations healthcare salaries based on time spend on treatment and transportation of medicatoin and/or patients through analysis of quantitative data

CONTACTS AND LOCATIONS:
Overall Officials: Karin Dieperink, RN, PhD, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenberg T, Kirkegaard J, Gundesen MT, Rasmussen MK, Dieperink KB, Lund T. Home-Based Daratumumab in Patients With Multiple Myeloma. Eur J Haematol. 2025 Jul;115(1):72-81. doi: 10.1111/ejh.14409. Epub 2025 Mar 31. PMID 40165411